CLINICAL TRIAL: NCT06000488
Title: Open-label Controlled Trial to Evaluate the Efficacy of a Manualized Reflective Writing Program for Clinical Phase PA Students.
Brief Title: Trial to Evaluate the Efficacy of a Manualized Reflective Writing Program for Clinical Phase Physician Assistant (PA) Students.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Yale PI left institution
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000035615
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Burn Out; Student Burnout; Physician Assistant Student Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The study sample will consist of clinical-phase PA students enrolled in the Yale Physician Associate Program Class of 2024.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention
- Reflective Writing Workshop Sessions (RWW) (Experimental): Participants will participate in three 75-minute RWW sessions scheduled to take place after students finish their 1st, 3rd, and 5th clinical rotations during the study period. reflective writing workshops
  Interventions: Behavioral: Reflective Writing Workshop Sessions

INTERVENTIONS:
Behavioral: Reflective Writing Workshop Sessions — Three workshops of 75 minutes. Trained PA and/or MD student facilitators will then use prepared materials to guide each group through a series of prompts, each eliciting written reflections of varying lengths. While all participants are encouraged to reflect, write, and share their responses, participation at all levels remains optional.
  Arms: Reflective Writing Workshop Sessions (RWW)

SUMMARY:
The following will be an open label controlled efficacy trial of the effects of longitudinal participation in an existing reflective writing program for medical students on burnout in physician assistant students.

DETAILED DESCRIPTION:
The pilot of the reflective writing workshop for PA students will follow the existing curriculum used for the MD program. The workshops will run for 75 minutes with additional time at the end of the session to complete a post-intervention assessment survey. Planning and adaptation of the program materials will be conducted by a group of PA students and the current MD-student leaders of the reflective writing program under the guidance of Dr. Anna Reisman.

All PA student participants will be split up into 1-2 groups of 6-10 students based on the number of participants. Sessions are expected to be held in-person pending COVID-19 guidance and will be held in reserved classroom space in the PA program building (100 Church Street South) or in reserved conference rooms at the Cushing-Whitney Medical Library. Trained PA and/or MD student facilitators will then use prepared materials to guide each group through a series of prompts, each eliciting written reflections of varying lengths. While all participants are encouraged to reflect, write, and share their responses, participation at all levels remains optional. Facilitators will not solicit any participants for a response. All program participants will be asked to complete a brief post-assessment survey consisting of short-answer and Likert scale questions about their attitudes towards program participation. Responses collected will be used to assess the feasibility and acceptability of the program for PA students and as feedback to guide potential future implementation of the program.

ELIGIBILITY:
Inclusion Criteria:

* able to offer consent
* able to speak and read English.
* must be a student in Yale Physician Associate Program Class of 2024

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in total burnout score over time as measured by the Copenhagen Burnout Inventory (CBI) | baseline (week 0), and weeks 4,12, and 26
  The Copenhagen Burnout Inventory (CBI) is a well-validated 19-item questionnaire used to measure burnout in different groups (e.g. employees, medical trainees, students) across three domains (personal, work, and client/customer). Total scores range from 0 to 100. Higher scores are associated with greater levels of burnout.

SECONDARY OUTCOMES:
Attitudes and mediators of behavioral change assessed by self report | week 26
  Attitudes and potential mediators of behavioral change will be assessed using a post-assessment survey consisting of short-answer and Likert-scale questions to be answered only by individuals who complete the active intervention. The survey will be distributed and completed at the end of each reflective writing workshop session. Analysis of the short response questions will use a rapid qualitative analysis method to identify patterns and themes. Likert-scale data will be analyzed by calculating the percentage of responses selecting each of the 5 dichotomous answer choices. A mean total score will be calculated through summation of all Likert scale categories as a numeric variable from 1-5, with higher scores indicating more positive responses for each question (e.g. Completely agree = 5 pts).

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Chiang, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No